CLINICAL TRIAL: NCT03042429
Title: Combination Chemotherapy Followed by Stem Cell Transplant and Isotretinoin in Treating Young Patients With High-risk Neuroblastoma
Brief Title: Combination Chemotherapy Followed by Stem Cell Transplant in High-risk Neuroblastoma Patients
Acronym: NB2004-HR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Frank Berthold, Prof. Dr., University of Cologne
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UCologne
Record Dates: First submitted 2017-02-01; First posted 2017-02-03 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Neuroblastoma
Keywords: neuroblastoma; chemotherapy; autologous stem cell transplantation; radiotherapy; mIBG; tumor resection
MeSH Terms: conditions — Neuroblastoma | interventions — Topotecan; Cyclophosphamide; Etoposide; Cisplatin; Vindesine; Ifosfamide; Doxorubicin

STUDY DESIGN:
Intervention Model Description: Randomized, multi-center, non-blinded, prospective, controlled trial
Masking Description: no masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental arm (Experimental): Drug: Cycles N8, N5, and N6 Drug: topotecan, cyclophosphamide, and etoposide (N8 cycle) followed by Drug: cisplatin, etoposide, and vindesine (N5 cycle) and Drug: vincristine, dacarbacine, ifosfamide, and doxorubicine (N6 cycle) followed by myeloablative chemotherapy with autologous stem cell transplantation (melphalan, carboplatin, etoposide) and by 9 x retinoic acid cycles (6 months, 3 months break, 3 months)
  Interventions: Drug: Cycles N8, N5 and N6
- standard arm (Active Comparator): Drug: Cycles N5 and N6 Drug: cisplatin, etoposide, and vindesine (N5 cycle) and Drug: vincristine, dacarbacine, ifosfamide, and doxorubicine (N6 cycle) followed by myeloablative chemotherapy with autologous stem cell transplantation (melphalan, carboplatin, etoposide) and by 9 x retinoic acid cycles (6 months, 3 months break, 3 months)
  Interventions: Drug: Cycles N5 and N6

INTERVENTIONS:
Drug: Cycles N8, N5 and N6 — two chemotherapy cycles N8 followed by standard arm therapy
  Other Names: topotecan, cyclophosphamide, etoposide
  Arms: experimental arm
Drug: Cycles N5 and N6 — Standard arm six chemotherapy cycles (3xN5 and 3x N6) followed by myeloablative therapy with stem cell support and isotretinoin
  Other Names: cisplatin, vindesine, ifosfamide, dacarbacine, doxorubicine
  Arms: standard arm

SUMMARY:
Improvement of event free survival of high-risk neuroblastoma patients by introduction of two additional topotecan containing chemotherapy cycles into the multimodal standard treatment (induction chemotherapy, myeloablative therapy, radiation, surgery as indicated, and consolidation therapy).

DETAILED DESCRIPTION:
Experimental intervention (6 weeks + duration of the control intervention):

2 x N8 cycle (topotecan, cyclophosphamide, and etoposide) followed by standard arm treatment (i.e., control intervention)

Control intervention (total duration 70-76 weeks):

3 x N5 cycle (cisplatin, etoposide, and vindesine) 3 x N6 cycle (vincristine, dacarbacine, ifosfamide, and doxorubicine), myeloablative chemotherapy with autologous stem cell transplantation (melphalan, carboplatin, etoposide) 9 x retinoic acid cycles (6 months, 3 months break, 3 months) supportive care (PCP/fungal prophylaxis, transfusions, antibiotics, G-CSF)

ELIGIBILITY:
Inclusion Criteria:

* neuroblastoma
* stage 4 neuroblastoma and age ≥1 - 21 years or MYCN amplification and age ≥6 months - 21 years
* informed consent obtained

Exclusion Criteria:

* Participation in other trials
* Pregnancy, lactation, or insufficient contraception for girls in childbearing age,
* Any concomitant non-protocol anticancer therapy,
* Incomplete initial staging.

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 360 (Actual)
Dates: Start 2007-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Event free survival | up to 9 years
  days from diagnosis to Event or last follow-up

SECONDARY OUTCOMES:
Overall survival | up to 9 years
  days from diagnosis to death or last follow-up
early response | up to 3 months
  remission status (INRG) measured after 2 chemotherapy cycles
late response | up to 9 months
  remission status (INRG) measured before stem cell transplant

CONTACTS AND LOCATIONS:
Overall Officials: Frank Berthold, Prof., Study Chair — University of Cologne
Locations (1):
- University of Cologne, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Berthold F, Hero B, Kremens B, Handgretinger R, Henze G, Schilling FH, Schrappe M, Simon T, Spix C. Long-term results and risk profiles of patients in five consecutive trials (1979-1997) with stage 4 neuroblastoma over 1 year of age. Cancer Lett. 2003 Jul 18;197(1-2):11-7. doi: 10.1016/s0304-3835(03)00076-4. PMID 12880954
- [Result] Berthold F, Boos J, Burdach S, Erttmann R, Henze G, Hermann J, Klingebiel T, Kremens B, Schilling FH, Schrappe M, Simon T, Hero B. Myeloablative megatherapy with autologous stem-cell rescue versus oral maintenance chemotherapy as consolidation treatment in patients with high-risk neuroblastoma: a randomised controlled trial. Lancet Oncol. 2005 Sep;6(9):649-58. doi: 10.1016/S1470-2045(05)70291-6. PMID 16129365
- [Result] Langler A, Christaras A, Abshagen K, Krauth K, Hero B, Berthold F. Topotecan in the treatment of refractory neuroblastoma and other malignant tumors in childhood - a phase-II-study. Klin Padiatr. 2002 Jul-Aug;214(4):153-6. doi: 10.1055/s-2002-33175. PMID 12165894
- [Result] Berthold F, Hero B. Neuroblastoma: current drug therapy recommendations as part of the total treatment approach. Drugs. 2000 Jun;59(6):1261-77. doi: 10.2165/00003495-200059060-00006. PMID 10882162